CLINICAL TRIAL: NCT06241872
Title: Evaluation of the Effectiveness of Dry Needling Treatment in Patients Diagnosed with Greater Trochanteric Pain Syndrome Accompanied by Myofascial Pain Syndrome
Brief Title: Evaluation of the Effectiveness of Dry Needling Treatment in Patients Diagnosed with Greater Trochanteric Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hasan Hüseyin Gökpınar, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KutahyaHSU-DRGOKPINAR-43
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Greater Trochanteric Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry needling group (study group) (Experimental): For patients in this group, dry needling will be performed once a week for three weeks on trigger points described as pain points in the Copeman nodule, gluteus medius, gluteus maximus, and iliotibial band muscles, guided by ultrasound. Patients will be instructed to perform daily stretching exercises outlined in the home program and mark their daily use of paracetamol on the provided schedule if needed. They will refrain from using NSAIDs or steroids during this period.
  Interventions: Other: Dry needling group
- Sham dry needling group (control group) (Sham Comparator): For the patients in this group, dry needling will be performed once a week for three weeks on trigger points described as pain points in the Copeman nodule, gluteus medius, gluteus maximus, and iliotibial band muscles, guided by ultrasound. However, the needles will not penetrate beyond the subcutaneous fatty tissue. Patients will be instructed to perform daily stretching exercises outlined in the home program and mark their daily use of paracetamol on the provided schedule if needed. They will refrain from using NSAIDs or steroids during this period.
  Interventions: Other: Dry needling group

INTERVENTIONS:
Other: Dry needling group — Dry needling will be performed using a 27-gauge, 5 cm long dental needle, guided by ultrasound, on predetermined trigger points in patients.
  Other Names: Study group

SUMMARY:
Greater Trochanteric Pain Syndrome (GTPS) is characterized by lateral hip pain, pain radiating to the lateral leg, tenderness and rotation around the greater trochanter, and pain with specific activities such as abduction or adduction. GTPS is primarily diagnosed clinically. Conservative treatment for GTPS includes activity modification, physiotherapy, nonsteroidal anti-inflammatory drugs, local corticosteroids, and platelet-rich plasma injections. Particularly, regional muscle sensitivity, such as in the gluteus maximus, is prominent. In recent years, dry needling therapy, which has gained popularity and increased research attention, has become an alternative treatment option, especially if the underlying cause is myofascial pain syndrome or deeper issues like piriformis syndrome.

The provided text discusses dry needling as a treatment for various neuromusculoskeletal pain conditions, emphasizing its use as a minimally invasive procedure that involves applying filiform needles to the relevant muscle tissue without the administration of pharmacological drugs. The literature suggests that dry needling therapy has the ability to induce biochemical, biomechanical, endocrinological, and neurovascular changes associated with the reduction of pain and disability in individuals. However, the optimal treatment dosage has not yet been determined, and there is inconsistency in the literature regarding the number of needles to be inserted and the duration of needle retention.

Studies evaluating the effectiveness of dry needling are often designed to compare or add it to other injection therapies. Additionally, there is a limited number of studies conducted with real-time imaging. In the planned study, the use of ultrasound-guided dry needling aims to provide a sham application opportunity, where the patient is blinded to the nature of the procedure, allowing for a meaningful investigation of efficacy. This aspect of the study is expected to contribute significantly to the literature.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 80 years old. Ability to read and write. Clinically diagnosed with greater trochanteric pain syndrome. Pain Visual Analog Scale (VAS) score of 6 or higher.

Exclusion Criteria:

History of previous lumbar and hip surgery. Lesions, atrophy, or scars in the skin around the hip area. Received physiotherapy for the hip, lumbar, or lower extremities in the last 6 months.

Underwent an interventional procedure for the hip or lumbar region for the same reason in the last 3 months.

Used steroids in the last 1 month. Special conditions such as epilepsy, pregnancy, injection phobia, etc. Inability to comply with the restriction on the use of both steroid and non-steroidal anti-inflammatory drugs during the treatment period.

Subcutaneous fat tissue thickness in the hip area being 5 cm or more.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: Up to 24 hour before the third intervention, Time frame 4: One week (and one month) after the last intervention.
  "Visual Analog Scale (VAS)" is a measurement instrument often used in healthcare to assess the intensity or characteristics of subjective experiences such as pain. It typically consists of a straight line, usually 10 centimeters in length, with endpoints representing extremes (e.g., "no pain" to "worst imaginable pain"). Patients mark on the line to indicate their subjective experience, and the distance from one endpoint provides a numerical score representing the intensity of the sensation being measured. The VAS is commonly employed in pain assessment but can also be adapted for various other subjective evaluations.
Patient-Specific Functional Scale | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: Up to 24 hour before the third intervention, Time frame 4: One week (and one month) after the last intervention.
  "Patient-Specific Functional Scale" (PSFS). The PSFS is a self-report outcome measure commonly used in healthcare, particularly in physical therapy and rehabilitation settings. It is designed to assess the patient's perceived difficulty in performing specific activities that are relevant to their daily life and function. Identification of Activities: The patient is asked to identify and list three to five activities that they find challenging or have difficulty performing due to their condition or symptoms.
  Rating Scale: For each identified activity, the patient is asked to rate their current level of difficulty on a numerical scale, often ranging from 0 to 10. A score of 0 indicates no difficulty, while 10 indicates the maximum difficulty.
  Follow-up Assessments: The same activities and rating scale are used in follow-up assessments to track changes over time or in response to interventions.

SECONDARY OUTCOMES:
Pressure Pain Threshold Measurement | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: Up to 24 hour before the third intervention, Time frame 4: One week (and one month) after the last intervention.
  "Pressure Pain Threshold Measurement" refers to the assessment of the amount of pressure applied to a specific point on the body before the individual perceives it as painful. This measurement is commonly used in clinical settings to evaluate pain sensitivity and threshold. The process involves gradually applying pressure to a specific area until the individual signals that they begin to feel pain. It is a quantitative way to assess pain perception and is often utilized in research, physical therapy, and other healthcare disciplines to understand pain levels and responses.
The Oswestry Disability Index | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention.
  Oswestry Disability Index (ODI) specifically designed to assess the impact of low back pain on a person's daily activities and functioning. The Oswestry Disability Index is a widely used self-report questionnaire that helps quantify the degree of disability experienced by individuals with low back pain.The ODI typically consists of ten sections, each addressing a different aspect of daily life and function. The sections cover topics such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment or other daily activities. For each section, individuals rate their level of disability, and the overall score is calculated as a percentage of the maximum possible disability.
Hip ROM Measurement | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention.
  Range of motion (ROM) in the hip joint is a crucial aspect of musculoskeletal function, and measuring it can provide valuable information about joint health, flexibility, and potential issues related to the hip.
  Hip ROM measurements typically involve assessing the movement capabilities of the hip joint in different directions, including flexion, extension, abduction, adduction, internal rotation, and external rotation

CONTACTS AND LOCATIONS:
Overall Officials: Hasan H Gökpınar, Ass. Prof., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No